CLINICAL TRIAL: NCT06542016
Title: A Prospective Study on Predicting Cardiovascular Events and Mortality Risk in Maintenance Dialysis Patients Based on Changes in KCCQ Scores
Brief Title: An Evaluation of the KCCQ Score in Predicting Cardiovascular Risk in Dialysis Patients
Status: Recruiting | Type: Observational
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Xu, Principal Investigator, Shenzhen Second People's Hospital
Other Study IDs: 20240625123
Record Dates: First submitted 2024-07-30; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Disease Stage 5; Dialysis; Heart Failure
Keywords: Chronic Kidney Disease Stage 5; Maintenance Dialysis; Heart Failure; Cardiovascular Outcomes; Kansas City Cardiomyopathy Questionnaire; patient self-reported outcomes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular Disease (CVD) is the main complication and the most important cause of death in CKD patients. As the disease progresses, the incidence of cardiovascular disease in CKD patients gradually increases, especially in End-Stage Renal Disease (ESRD) patients receiving dialysis treatment, where the prevalence of cardiovascular disease reaches its highest level. Currently, there is a lack of a simple and reliable tool to assess the cardiac function status and predict the risk of cardiovascular events in patients on maintenance dialysis. The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a widely used patient-reported outcomes measurement tool for assessing health-related quality of life in heart failure patients. It has been shown that KCCQ scores not only reflect the underlying undiagnosed symptoms of heart failure in CKD patients, but also have a strong correlation with prognosis. However, there is currently insufficient clinical evidence to confirm the value of the KCCQ in patients on maintenance dialysis.

Investigators will perform a prospective, single-center, observational study to collect the changing trend of KCCQ scores at baseline and during the observation periods in maintenance dialysis patients, to analyze the association between the scores and the occurrence of long-term cardiovascular events and all-cause mortality. The aim is to construct a predictive model of KCCQ scores to provide a reference basis for clinical management of this high-risk group, so as to optimize the diagnosis and treatment of heart failure in dialysis patients and improve their cardiovascular outcomes.

DETAILED DESCRIPTION:
Investigators will apply the KCCQ to maintenance dialysis patients and statistically analyze baseline KCCQ scores and changing trends to investigate whether they are associated with the occurrence of long-term cardiovascular events and all-cause mortality in dialysis patients and to construct a predictive model associated with KCCQ scores. Patients who meet the inclusion and exclusion criteria will sign an informed consent form, and the baseline index test and the KCCQ assessment will be performed within one week after enrollment. Then the follow-up will be conducted according to the follow-up plan (KCCQ scores and test indexes will be collected at 0, 1, 2, 3, 6, 9 and 12 months in patients with new-onset uremia and the patients with maintenance dialysis will be collected at 0, 3, 6, 9 and 12 months). Conduct a KCCQ assessment and collect relevant indicators during each follow-up visit. There is no intervention in the patient's treatment regimen during the study period. All participants enrolled in the study will be followed up for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older with no restrictions on gender or ethnicity;
2. All enrolled patients meet the diagnostic criteria for CKD stage 5 according to the KDOQI guidelines of the National Kidney Foundation;
3. Newly diagnosed uremia patients planning to start maintenance dialysis (hemodialysis or peritoneal dialysis), as well as patients currently undergoing maintenance dialysis treatment (hemodialysis or peritoneal dialysis);
4. Clear contact information is available to reach patients or family members for follow-up;
5. Signed informed consent and ability to complete the KCCQ.

Exclusion Criteria:

1. Patients with acute kidney injury from various causes;
2. Patients with severe mental illnesses that affect their ability to complete questionnaires;
3. Patients who have had acute myocardial infarction, coronary artery stent implantation, coronary artery bypass grafting (CABG) or pacemaker implantation within the past three months;
4. Patients with special types of heart disease, including cardiac amyloidosis, congenital heart disease and pericardial diseases;
5. Patients with chronic lung diseases;
6. Patients with serious underlying conditions such as severe infections, tumors or severe liver diseases;
7. Patients scheduled for kidney transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll at least 136 patients meeting inclusion and exclusion criteria who are either currently undergoing maintenance dialysis or newly diagnosed with uremia and scheduled to start maintenance dialysis from July to December 2024 in the Nephrology Department of Shenzhen Second People's Hospital. The study will follow these patients for at least 12 months. During this period, the KCCQ scores and relevant test indicators will be collected regularly to explore the relationship between the baseline KCCQ scores and changes in scores and the occurrence of long-term cardiovascular events and all-cause mortality.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 12 months
  All-cause mortality is defined as death from any cause during the study period. This primary outcome measure will assess the occurrence of death among study participants, regardless of the specific cause.
Mortality from cardiovascular causes | 12 months
  Mortality from cardiovascular causes includes deaths resulting from conditions such as myocardial infarction, heart failure, stroke and other cardiovascular event. This primary outcome measure will assess deaths specifically attributed to cardiovascular causes among study participants.
Incidence of cardiovascular disease-related hospitalizations | 12 months
  Cardiovascular disease-related hospitalizations include admissions for conditions such as acute coronary syndrome, heart failure exacerbation, stroke, arrhythmias and other cardiovascular events requiring inpatient care. The primary outcome measure will assess the occurrence of hospitalizations related to cardiovascular diseases among study participants.

CONTACTS AND LOCATIONS:
Overall Officials: QiJun Wan, Study Director — Shenzhen Second People's Hospital
Locations (1):
- First Shenzhen, Guangdong, Guangdong, China